CLINICAL TRIAL: NCT03820817
Title: Pilot Study of Oral Rifaximin in Patients With Monoclonal Gammopathy
Brief Title: Rifaximin in Patients With Monoclonal Gammopathy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106380; NCI-2018-02106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4480-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: IgA Monoclonal Gammopathy; IgG Monoclonal Gammopathy; IgM Monoclonal Gammopathy; Light Chain Deposition Disease; Monoclonal Gammopathy; Smoldering Waldenstrom Macroglobulinemia; Waldenstrom Macroglobulinemia; Gammopathy, Monoclonal; Gammopathy Igg
MeSH Terms: conditions — Paraproteinemias; Waldenstrom Macroglobulinemia | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rifaximin) (Experimental): Patients receive rifaximin PO TID on days 1-14 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Given PO
  Other Names: Xifaxan

SUMMARY:
This trial studies how well rifaximin works in treating patients with monoclonal gammopathy. Antibiotics, such as rifaximin, may help to kill bacteria in the intestines and reduce the abnormal protein or cells in patients with monoclonal gammopathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of a 2-week course of rifaximin on clonal immunoglobulin (Ig) in patients with monoclonal gammopathy.

SECONDARY OBJECTIVES:

I. To evaluate safety and tolerability of a 2-week course of rifaximin.

II. To evaluate changes in stool microbiota by 16S ribosomal ribonucleic acid (rRNA) gene (16S) sequencing.

III. To evaluate changes in gammopathy as assessed by changes in clonal Ig and/or plasma cells.

OUTLINE:

Patients receive rifaximin orally (PO) thrice daily (TID) on days 1-14 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of monoclonal gammopathy of undetermined significance based on International Myeloma Working Group (IMWG) criteria
* Patients will be enrolled into one of 3 cohorts:

  * Cohort A: IgA gammopathy
  * Cohort B: IgG gammopathy / or light chain gammopathy
  * Cohort C: IgM gammopathy / asymptomatic macroglobulinemia
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received antibiotics within last 3 weeks
* Patients who are receiving any other investigational agents for gammopathy. Patients with clinical myeloma requiring anti-myeloma therapy are also excluded
* History of allergic reactions or intolerance attributed to rifaximin or compounds of similar chemical or biologic composition to antibiotic under study
* The effects of rifaximin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of rifaximin administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate defined as a reduction in clonal immunoglobulin (Ig) by > 25% | Up to 2 weeks after study start
  Clinical response rate will be calculated as proportion (responders/total patients).

SECONDARY OUTCOMES:
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 12 weeks after study start
  Incidence of adverse events (AEs) occurring during the study will be summarized by system organ class and preferred term. Adverse events will also be summarized by causality and grade. Serious adverse events will be listed separately.
Changes in stool microbiota | Up to 12 weeks after study start
  16S sequencing will be used to compare changes in stool microbiota.
Changes in gammopathy | Up to 12 weeks after study start
  Changes in clonal Ig will be used to assess changes in gammopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Nooka, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No